CLINICAL TRIAL: NCT03141723
Title: Randomized Trials of Kangaroo Mother Care With Plastic Bag to Prevent Neonatal Hypothermia in Preterm Infants (Trial 2A and 2B)
Brief Title: Kangaroo Mother Care With Plastic Bag (Trials 2A & 2B)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other)
Responsible Party: Principal Investigator, Colm Travers, MD, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F150807003
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Preterm Infant; Hypothermia Neonatal
Keywords: Infant; Newborn; Preterm; Hypothermia; Kangaroo; Plastic; Bag
MeSH Terms: conditions — Premature Birth; Hypothermia

STUDY DESIGN:
Intervention Model Description: Randomization at birth followed by randomization at 1 hour
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KMC & WHO protocol (0-1 hour) (Active Comparator): The combination of Kangaroo Mother Care (KMC) as continuously as possible together with routine World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling.
  Interventions: Other: KMC & WHO protocol (0-1 hour)
- KMC & WHO protocol (1-24 hours) (Active Comparator): The combination of Kangaroo Mother Care (KMC) as continuously as possible together with routine World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling.
  Interventions: Other: KMC & WHO protocol (1-24 hours)
- KMC, WHO protocol & bag (0-1 hour) (Experimental): The combination of Kangaroo Mother Care (KMC) as continuously as possible together with the use of a plastic bag in combination with routine World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling.
  Interventions: Other: KMC, WHO protocol & bag (0-1 hour)
- KMC, WHO protocol & bag (1-24 hours (Experimental): The combination of Kangaroo Mother Care (KMC) as continuously as possible together with the use of a plastic bag in combination with routine World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling.
  Interventions: Other: KMC, WHO protocol & bag (1-24 hours)

INTERVENTIONS:
Other: KMC & WHO protocol (0-1 hour) — WHO thermoregulation care - warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling.
  Arms: KMC & WHO protocol (0-1 hour)
Other: KMC, WHO protocol & bag (0-1 hour) — In addition infants will be placed in a plastic bag (clear polyethylene nonmedical low-cost [3 cents per bag] linear low-density bag measuring 10 × 8 × 24 in. and 1.2 mil thick) that will cover the infant's torso and lower extremities.
  Arms: KMC, WHO protocol & bag (0-1 hour)
Other: KMC & WHO protocol (1-24 hours) — WHO thermoregulation care - warm delivery rooms, immediate drying after birth, early and exclusive
  Arms: KMC & WHO protocol (1-24 hours)
Other: KMC, WHO protocol & bag (1-24 hours) — In addition infants will be placed in a plastic bag (clear polyethylene nonmedical low-cost [3 cents per bag]
  Arms: KMC, WHO protocol & bag (1-24 hours

SUMMARY:
The purpose of this study is to determine whether the combination of Kangaroo Mother Care (KMC) as continuously as possible together with the use of a plastic bag in combination with routine World Health Organization (WHO) thermoregulation care reduces the incidence of moderate (32-36° C) or severe (<32.0° C) hypothermia in term infants ≥ 37 0/7 weeks of gestational age (GA) when compared to KMC as continuously as possible together with routine WHO thermoregulation care.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the combination of Kangaroo Mother Care (KMC) as continuously as possible together with the use of a plastic bag in combination with routine World Health Organization (WHO) thermoregulation care (warm delivery rooms, immediate drying after birth, early and exclusive breastfeeding, postponement of bathing and weighing, and appropriate bundling) reduces the incidence of moderate hypothermia (32-36° C) or severe (<32.0° C) in term infants ≥ 37 0/7 weeks of gestational age (GA) when compared to KMC as continuously as possible together with routine WHO thermoregulation care, as practiced. The investigators are proposing two trials, one protocol for infants 32-36 6/7 weeks and one for infants who are ≥37 weeks gestational age (this one). This term infant trial will address the effectiveness of KMC in combination with plastic bags in decreasing hypothermia in preterm infants. The proposed trial will determine whether KMC with plastic bags prevents hypothermia in neonates born in a healthcare setting with limited resources where a high risk for hypothermia has been reported. Any intervention that decreases morbidity during the neonatal period has the potential to impact health beyond the neonatal period,and one that is highly cost-effective and easy to use is more likely to be implemented in the developing world.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age ≥37 0/7 weeks
* Delivery in the hospital

Exclusion Criteria:

* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder
* Clinically unstable mothers secondary to cardiovascular and pulmonary conditions
* Infants requiring respiratory support beyond 10 minutes after birth
* Infant requiring Neonatal Intensive Care Unit admission
* Cesarean section
* Multiple gestation if the last delivering infant is not born within 10 minutes from the time of birth of the first infant

Ages: 10 Minutes to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 423 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2017-08-12 (Actual)

PRIMARY OUTCOMES:
Moderate or severe hypothermia at 1 hour after birth (Phase 2A) | 1 hour after birth
  Moderate (32.0-35.9C) or severe (<32.0C) hypothermia at 1 hour after birth (via axillary temperature)
Moderate or severe hypothermia at 24 hours or discharge (Phase 2B) | 1 to 24 hours after birth
  Moderate (32.0-35.9C) or severe (<32.0C) hypothermia at 24 hours or discharge whichever occurs first (via axillary temperature)

SECONDARY OUTCOMES:
Any hypothermia at 1 hour after birth (Phase 2A) | 1 hour after birth
  Any hypothermia (<36.5C) at 1 hour after birth
Any hypothermia at 1 hour after birth (Phase 2B) | 1 to 24 hours or discharge
  Any hypothermia (<36.5C) at 24 hours or discharge, whichever occurs first
Hyperthermia at 1 hour after birth (Phase 2A) | 1 hour after birth
  Hyperthermia (>38.0C) at 1 hour after birth
Hyperthermia at 1 hour after birth (Phase 2B) | 1 to 24 hours or discharge
  Hyperthermia (>38.0C) at 24 hours or discharge, whichever occurs first
Skin rash | 1 hour to 24 hours or discharge, or whichever occurs first
  Skin rash (at 1 hour and before discharge)
Neonatal Intensive Care Unit admission | 1 hour to 24 hours or discharge, or whichever occurs first
  Neonatal Intensive Care Unit admission (at 1 hour and before discharge)
Respiratory distress syndrome | 1 hour to 24 hours or discharge, or whichever occurs first
  Diagnosis of respiratory distress syndrome (at 1 hour and before discharge)
Sepsis | 1 hour to 24 hours or discharge, or whichever occurs first
  Diagnosis of sepsis (at 1 hour and before discharge)
Hypotension, hypoglycemia or seizure | 1 hour to 24 hours or discharge, or whichever occurs first
  Diagnosis of any of the following; hypotension, hypoglycemia or seizure (at 1hour and before discharge)
Death | 1 hour to 24 hours or discharge, or whichever occurs first
  Death (at 1 hour and before discharge)
Maternal body temperature | At birth, at 1 hour, and every four hours until 24 hours or discharge, whichever occurs first
  Maternal body temperature in Celsius
Duration of KMC and plastic bag to infant's body temperature | During first 1 hour
  Correlation analysis between duration of KMC +/- plastic bag in minutes to infant's body temperature in Celsius
Duration of KMC and plastic bag to infant's body temperature | During first 24 hours or discharge, or whichever occurs first]
  Correlation analysis between duration of KMC +/- plastic bag in minutes to infant's body temperature in Celsius

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, MD, Principal Investigator — University of Alabama at Birmingham; Waldemar A Carlo, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travers CP, Ramani M, Gentle SJ, Schuyler A, Brown C, Dills MM, Davis CB, Mwenechanya M, Chomba E, Aban I, Manasyan A, Ambalavanan N, Carlo WA. Early Skin-to-Skin Care with a Polyethylene Bag for Neonatal Hypothermia: A Randomized Clinical Trial. J Pediatr. 2021 Apr;231:55-60.e1. doi: 10.1016/j.jpeds.2020.12.064. Epub 2020 Dec 26. PMID 33373672